CLINICAL TRIAL: NCT06145750
Title: Implementing Fragmentomics Into Real World Screening IntervenTions to Evaluate Clinical Utility Among Individuals With Elevated Risk for Lung Cancer
Acronym: FIRSTLUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delfi Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DELFI-L301
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Lung Cancer Screening; Early Diagnosis; Low Dose CT Scan; CT Scan; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Lung Diseases; Respiratory Tract Diseases; Biomarkers; Lung Cancer Prevention; Fragmentomics; CAT Scan; Early Detection; NSCLC; Adenocarcinoma; Lung Malignancy; Liquid Biopsy; LDCT
MeSH Terms: conditions — Lung Neoplasms; Disease; Respiratory Tract Neoplasms; Thoracic Neoplasms; Lung Diseases; Respiratory Tract Diseases; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Physician practices (the study participants) will be randomized 1:1:2 to Arm A1 (control), Arm A2 (Control) or Arm B (intervention). Arm A practices will be further randomized 1:1 into two groups (A1:A2) to observe lung cancer screening standard of care. Practices in A1 will be observed; practices in A2 will receive standard education on lung cancer screening for Continuing Medical Education (CME) credit. Randomizing within Arm A aims to delineate the impact standard lung cancer screening education may have on utilization. Arm B (intervention) practices will receive education on FirstLook™ and have access to order FirstLook™ at the providers' discretion. A limited data set (LDS) will be extracted from the primary care practice EMRs for the study analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A1 (No Intervention): Arm A practices will be further randomized 1:1 into two groups (A1:A2) to observe lung cancer screening standard of care. Practices in A1 will be observed.
- Arm A2 (Active Comparator): Arm A practices will be further randomized 1:1 into two groups (A1:A2) to observe lung cancer screening standard of care. Practices in A2 will receive standard education on lung cancer screening for CME credit.
  Interventions: Other: Continuing Medical Education for Lung Cancer
- Arm B (Experimental): Arm B (intervention) practices will receive education on FirstLook™ and have access to order FirstLook™ at the providers' discretion;
  Interventions: Diagnostic Test: Ability to order FirstLook™

INTERVENTIONS:
Diagnostic Test: Ability to order FirstLook™ — FirstLook™ is a commercially available, validated next generation sequencing assay of plasma cell-free DNA (cfDNA) that analyzes the distribution of cfDNA fragment sizes to indicate the presence of possible lung cancer. FirstLook™ is intended to be used by a qualified healthcare provider and is not a replacement for computed tomography (CT) or low-dose computed tomography (LDCT). FirstLook™ is validated for use in individuals aged 50 to 80 who either currently or previously smoked cigarettes and accumulated 20 pack-years or more of exposure.
  Other Names: FirstLook™
  Arms: Arm B
Other: Continuing Medical Education for Lung Cancer — Physician practice will receive standard education on lung cancer screening for CME credit.
  Arms: Arm A2

SUMMARY:
The purpose of this study is to determine whether availability of DNA Evaluation of Fragments for Early Interception (DELFI) Lung Cancer Screening Test, FirstLook™ to practicing physicians affects overall lung cancer screening rates among their patients who are recommended and eligible for screening based on 2021 United States Preventive Services Task Force (USPSTF) but are not up to date with it. DELFI hypothesized that patients in the care of physicians or practice groups who have FirstLook™ will have increased lung screening rates compared to patients in the care of physicians or practice groups who do not have access to FirstLook™.

DETAILED DESCRIPTION:
Despite compelling evidence of the benefits of lung cancer screening, rates among eligible individuals in the United States remain stubbornly low. Using a cluster randomized controlled trial, DELFI plans to evaluate whether lung screening rates can be increased if physicians and practice groups have the ability to order a validated, commercially available FirstLook™ as an initial test for eligible individuals who are not up to date with lung screening recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Practice offers primary care services. Primary care services may include, but are not limited to: community health centers, academic outpatient facilities, private practices of family or general internal medicine, and Veterans Administration outpatient primary care clinics.
2. Practice has a lung cancer screening population of a minimum of 50 individuals upon first review of patient records. a. Lung cancer screening eligible population is defined as meeting the 2021 USPSTF guideline recommendations (current and former smokers 50-80 years of age, 20 pack year or more smoking history, have not quit more than 15 years ago) b. Individuals have had a clinic visit in the past 12 months, and c. Individuals have not had a CT for lung cancer screening in the last 15 months.
3. Practice can complete EMR data extraction and EDC entry during the study.
4. Practice scores a 4 (agree) or 5 (strongly agree) on a 5-point Likert scale for physical and payer benefit access to LDCT.
5. The practice utilizes conveniently located phlebotomy that accepts same-day services.

Exclusion Criteria:

1. Practice is currently participating in other DELFI studies.
2. Practice is actively participating in any other cancer screening blood-based biomarker studies which includes return of results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of practice-identified lung cancer screen-eligible individuals receiving any screening event, defined as either a screening CT (LDCT or chest CT) or FirstLook™ Lung test (FLL) blood draw during the study period in each arm. | 15 months

SECONDARY OUTCOMES:
Proportion of practice-identified lung cancer screen-eligible individuals receiving a screening CT scan during the study period in each arm. | 15 months
Proportion of practice-identified lung cancer screen-eligible individuals receiving a CT order and/or completed CT scan for lung cancer screening following FirstLook™ test result during the study period. | 15 months
Number needed to screen (NNS) with FirstLook™ to detect one additional lung cancer during the study period. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bach, MD, Study Chair — Chief Medical Officer
Locations (3):
- United States (3):
  - DARTNet Institute, Aurora, Colorado
  - University Of Florida, Jacksonville, Florida
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Detection and characterization of lung cancer using cell-free DNA fragmentomes — https://www.nature.com/articles/s41467-021-24994-w
- See also: Screening for Lung Cancer: CHEST Guideline and Expert Panel Report — https://pubmed.ncbi.nlm.nih.gov/34270968/
- See also: Genome-wide cell-free DNA fragmentation in patients with cancer — https://www.nature.com/articles/s41586-019-1272-6